CLINICAL TRIAL: NCT06492928
Title: Evaluation of Attentionnal Performance by PVT of Health Workers During Their Shift in Emergency Department
Brief Title: Attentionnal Performance of Shift Health Workers in Emergency Department
Acronym: Emerg-APoSHeW
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Roubaix (Other)
Collaborators: Boulogne sur Mer Hospital Center (Other); Centre Hospitalier de l'Arrondissement de Montreuil-sur-mer (Unknown); Centre Hospitalier Saint-Omer (Unknown); Centre Hospitalier de Bethune (Network); Centre Hospitalier de Lens (Other); Polyclinique de la Clarence (Unknown); Centre hospitalier de Dunkerque (Unknown); Centre Hospitalier de Douai (Other); Centre Hospitalier de Valenciennes (Network); Centre Hospitalier d'Hazebrouck (Unknown); Centre Hospitalier de Watrelos (Unknown); Centre Hospitalier de Denain (Unknown); Tourcoing Hospital (Other); GHICL (Unknown); Polyclinique de Grande Synthe (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-015
Record Dates: First submitted 2024-06-25; First posted 2024-07-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Work-Related Condition
Keywords: shift-work; PVT; Health worker; Attentionnal performance; Emergency department
MeSH Terms: conditions — Emergencies | interventions — Maslach Burnout Inventory; Perceived Stress Scale

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Psychomotor Vigilance Task — T0 - at the start of the shift: completion of the 1st PVT / socio-demographic and workstation questionnaire T1 - at the end of the shift: completion of the second PVT and questionnaire on the course of the shift that has just taken place T2 - 1 week after the end of the shift: additional questionnaire sent with scales to assess work-related fatigue (MBI), anxiety (PSS), sleep quality (PSQI) and chronotype (MEQ).
  Other Names: Maslach Burnout Inventory; Perceived Stress Scale; Pittsburgh Sleep Quality Index; Morningness-Eveningness Questionary

SUMMARY:
Atypical working hours can be a risk factor for workers. In fact, the body is subject to a circadian rhythm, which affects numerous physiological activities. These biological rhythms reflect the need for certain physiological activities to occur at a specific time of day. This cycle can be disrupted and shifted by external factors. This disruption of biological rhythms can manifest itself in the appearance of health effects.

The innovative nature of our work lies in the search for an alteration in psychomotor functions in nursing staff (subject to atypical working hours). To this end, we decided to study the concentration of care workers using a reflex-based psychomotor test, the Psychomotor Vigilance Test (PVT). Other factors will be studied in order to assess the factors that may affect this test.

DETAILED DESCRIPTION:
Population : All care staff in the emergency departments of the participating hospitals: physicians, residents, nurses and nursing assistants.

The main objective is to evaluate concentration in medical/non-medical staff at the start and end of a work shift.

To this end, we will evaluate the Psychomotor Vigilance Test (PVT) and its variation at the start and end of a shift in these personnel.

The endpoint is the difference in reflex time to a visual stimulus performed at the beginning and end of the shift with a 3-minute PVT Test.

The first secondary objective is to analyze the number of PVT errors. The criterion defining an error is a reaction time greater than 500ms.

The second secondary objective is to compare the PVT and its variation in certain subgroups. The subgroups compared will be defined according to the following criteria :

* Shift duration: Non-medical staff (<10h, >10h), Medical staff (6 to 10h, 10 to 15h, 15 to 24h) Staggered shift: start before 6h or end after 22h,
* Type of service: acute care, MCO, SSR (or emergency sector)
* Sleep quality (Pittsburgh Sleep Quality Index),
* Professional fatigue (Maslach Burnout lnventory),
* Anxiety (French official version of the PSS-14),
* Chronotype (Morningness-Eveningness Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Physicians,
* residents,
* nurses,
* nursing assistants

Exclusion Criteria:

* Students,
* paramedics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Health Workers who start their shift during the study duration
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of concentration in medical/non-medical staff at the start and end of a work shift. | Day 1
  To this end, we will evaluate the Psychomotor Vigilance Test (PVT) and its variation at the start and end of a shift in these personnel.
  The endpoint is the difference in reflex time to a visual stimulus performed at the beginning and end of the shift with a 3-minute PVT Test.

SECONDARY OUTCOMES:
The first secondary objective is to analyze the number of PVT errors. | Day 1
  The criterion defining an error is a reaction time greater than 500ms.
Sub-group analysis | Day 7
  The second secondary objective is to compare the PVT and its variation in certain subgroups. The subgroups compared will be defined according to the following criteria Shift duration: Non-medical staff (<10h, >10h), Medical staff (6 to 10h, 10 to 15h, 15 to 24h) Staggered shift: start before 6h or end after 22h, Type of service: acute care, MCO, SSR (or emergency sector) Sleep quality (Pittsburgh Sleep Quality Index), Professional fatigue (Maslach Burnout lnventory), Anxiety (French official version of the PSS-14), Chronotype (Morningness-Eveningness Questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Remy Diesnis, MD, Principal Investigator — Centre Hospitalier de Roubaix
Locations (4):
- France (4):
  - Emergency Department, General Hospital, Armentières, Nord
  - Emergency Department, General Hospital, Hazebrouck, Nord
  - Emergency Department, GHICL Saint-Philibert, Lomme, Nord
  - Emergency Department, General Hospital, Tourcoing, Nord

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agence nationale de sécurité sanitaire de l'alimentation, de l'environnement et du travail.; 2016 juin. Report No.: 2011-SA-0088.
- [Background] Thun E, Bjorvatn B, Torsheim T, Moen BE, Magerøy N, Pallesen S. Night work and symptoms of anxiety and depression among nurses: A longitudinal study. Work Stress. 2 oct 2014;28(4):376 86.
- [Background] Folkard S, Tucker P. Shift work, safety and productivity. Occup Med (Lond). 2003 Mar;53(2):95-101. doi: 10.1093/occmed/kqg047. PMID 12637593